CLINICAL TRIAL: NCT00009711
Title: The Impact of Pediatric Marrow Transplantation on Late Pulmonary Function
Brief Title: Study of Lung Function in Children Who Have Undergone Bone Marrow Transplantation
Status: Completed | Type: Observational
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Other Study IDs: 1097.00; FHCRC-1097.00; NCI-G00-1911; CDR0000065808 (Registry Identifier: PDQ)
Record Dates: First submitted 2001-02-02; First posted 2003-01-27 (Estimated); Last update posted 2013-05-01 (Estimated); Status verified 2013-04

CONDITIONS: Long-term Effects Secondary to Cancer Therapy in Children; Pulmonary Complications
Keywords: long-term effects secondary to cancer therapy in children; pulmonary complications

INTERVENTIONS:
Procedure: management of therapy complications

SUMMARY:
RATIONALE: Assessing the long-term effects of bone marrow transplant on lung function in patients may improve the ability to plan treatment.

PURPOSE: This clinical trial studies lung function in pediatric patients who have undergone bone marrow transplant.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the delayed effects of bone marrow transplantation preparative regimens on pulmonary function in children surviving at least 5 years after transplantation for hematologic malignancy.
* Determine the relationship between pulmonary function and growth rates in these patients.
* Determine the effect of growth hormone treatment on pulmonary function in these patients.
* Determine the relationship between pulmonary function and age at time of transplantation in these patients.
* Determine the incidence and severity of restrictive pulmonary disease, and whether these factors vary with increasing time after transplantation in these patients.

OUTLINE: Patients undergo respiratory history, signs and symptoms assessment, pulmonary function tests (PFT) including spirometry, lung volumes, and diffusion, oxygen saturation by pulse oximetry, and height measurement.

Patients are assessed at 5-10 years, 10-15 years, and over 15 years after bone marrow transplantation. Patients with abnormal PFTs are assessed at more frequent intervals as clinically indicated.

PROJECTED ACCRUAL: Approximately 280 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Patients who have undergone bone marrow transplantation for hematologic malignancy at least 5 years ago

  * Disease-free survivors at least 6 years of age AND
  * Under 18 years of age at time of transplantation
* Received prior allogeneic, unrelated donor, syngeneic, or autologous bone marrow transplantation
* Able to perform pulmonary function tests

PATIENT CHARACTERISTICS:

Age:

* See Disease Characteristics

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics

Chemotherapy:

* Not specified

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* Any prior preparative regimen allowed

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 280 (Estimated)
Dates: Start 1996-03; Primary Completion 2004-08 (Actual); Study Completion 2005-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean E. Sanders, MD, Study Chair — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States